CLINICAL TRIAL: NCT05031715
Title: Effectiveness of the Assumption of a Berberine Phytosoma-based Supplement on the Hematic Values of Glucose in a Group of Patients With Altered Fasting Glucose
Brief Title: Berberine and Altered Fasting Glucose
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Azienda di Servizi alla Persona di Pavia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ID 0912/14122018
Record Dates: First submitted 2021-08-27; First posted 2021-09-02 (Actual); Last update posted 2022-03-03 (Actual); Status verified 2021-08

CONDITIONS: Glucose Metabolism Disorders
MeSH Terms: conditions — Glucose Metabolism Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dietary supplement (Experimental): Berberine Phytosome
  Interventions: Dietary Supplement: Berberine Phytosome

INTERVENTIONS:
Dietary Supplement: Berberine Phytosome — 2 tablets of 550 mg per day (1 before lunch and 1 before dinner)

SUMMARY:
The aim of the study was to evaluate the effectiveness of a food supplement, berberine phytosome, which contributes to the control of blood sugar and the improvement of insulin resistance.

ELIGIBILITY:
Inclusion Criteria:

* Fasting blood glucose range:100-125 mg/dl

Exclusion Criteria:

* Diabetes mellitus

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-03-02 (Actual); Primary Completion 2020-05-28 (Actual); Study Completion 2022-07-25 (Estimated)

PRIMARY OUTCOMES:
Changes on insulin resistance | Changes from baseline insulin resistance at 4 weeks and at 8 weeks
  Homeostasis Model Assessment (pt), for evaluate insulin resistance if > 2,4
Changes on carbohydrate profile | Changes from baseline carbohydrate profile at 4 weeks and at 8 weeks
  Fasting Glucose (mg/dl)
Changes on carbohydrate profile | Changes from baseline carbohydrate profile at 4 weeks and at 8 weeks
  Glycated hemoglobin (%)

SECONDARY OUTCOMES:
Changes on anthropometry | Changes from baseline anthropometry at 4 weeks and at 8 weeks
  Weight (Kg)
Changes on anthropometry | Changes from baseline anthropometry at 4 weeks and at 8 weeks
  Body Mass Index (Kg/m2)
Changes on anthropometry | Changes from baseline anthropometry at 4 weeks and at 8 weeks
  Waist circumference (cm)
Changes on body composition | Changes from baseline body composition at 4 weeks and at 8 weeks
  Fat mass (g), Fat Free Mass (g), Visceral Adipose Tissue (g)
Changes on lipid profile | Changes from baseline lipid profile at 4 weeks and at 8 weeks
  Total Cholesterol (mg/dl), High density lipoprotein Cholesterol (mg/dl), Low density lipoprotein Cholesterol (mg/dl), Triglycerides (mg/dl), Apolipoprotein A (mg/dl), Apolipoprotein B (mg/dl)
Changes on Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | Changes from baseline Incidence of Treatment-Emergent Adverse Events at 4 weeks and at 8 weeks
  Alanine aminotransferase (IU/l), Aspartate aminotransferase (IU/l)
Changes on Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | Changes from baseline Incidence of Treatment-Emergent Adverse Events at 4 weeks and at 8 weeks
  Gamma Glutamyl Transferase (U/l)
Changes on Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | Changes from baseline Incidence of Treatment-Emergent Adverse Events at 4 weeks and at 8 weeks
  Creatinine (mg/dl)
Changes on Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | Changes from baseline Incidence of Treatment-Emergent Adverse Events at 4 weeks and at 8 weeks
  Glomerural Filtrate Rate (ml/min)

CONTACTS AND LOCATIONS:
Overall Officials: Mariangela Rondanelli, Principal Investigator — Fondazione Casemiro Mondino
Locations (1):
- Mariangela Rondanelli, Pavia, Italy